CLINICAL TRIAL: NCT01814020
Title: An Open,Single-centre Pilot Study of Efficacy and Safety of Topical MOB015B in the Treatment of Distal Subungual Onychomycosis (DSO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Responsible Party: Sponsor
Other Study IDs: MOB015B/Final 30-Aug-2012
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2013-06

CONDITIONS: Distal Subungual Onychomycosis
Keywords: DSO

INTERVENTIONS:
Drug: MOB015B

SUMMARY:
Assess efficacy and safety of topical MOB015B, applied daily during 48 weeks, in adults with fungal nail infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. 18 - 70 years
3. DSO of at least one of the great toe(s) affecting 25 % to 75 % of the target nail.
4. Positive culture for dermatophytes (i.e. Trichophyton species; T. rubrum or T. mentagrophytes)
5. Signed written informed consent

Exclusion Criteria:

1. Proximal subungual onychomycosis.
2. DSO of both great toenails where involvement has extended into the proximal portion of the target nail (unaffected proximal nail is less than 2 mm)
3. "Spike" of onychomycosis extending to eponychium of the target nail
4. Presence of dermatophytoma (defined as demarcated and localised thick masses of fungal hyphae and necrotic keratin between the nail plate and nail bed) on the target nail
5. Other conditions than DSO known to cause abnormal nail appearance
6. Topical antifungal treatment of the nails within 1 month before screening
7. Systemic use of antifungal treatment within 3 months before screening
8. History or signs of peripheral circulatory insufficiency and/or diabetic neuropathy
9. Immunosuppression
10. Participation in another clinical trial with an investigational drug or device during the previous 4 weeks before screening
11. Known allergy to any of the tested treatment products
12. A pregnancy test indicating pregnancy in a woman of childbearing potential at screening (visit 1)
13. Pre-menopausal (last menstruation ≤ 1 year prior to screening) sexually active women who :

    * are pregnant or nursing
    * are not surgically sterile
    * are of child bearing potential and not practising an acceptable method of birth control, or does not plan to continue practising an acceptable method of birth control throughout the trial (acceptable methods include intrauterine devices (IUD), oral, implantable or injectable contraceptives, diaphragm or cervical cap with intravaginal spermicide, condom with intravaginal spermicide or vasectomised partner)

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with mycological cure of the target nail,defined as negative fungal culture and negative direct microscopy at 60 weeks. | At 60 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hudkliniken Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden